CLINICAL TRIAL: NCT00409331
Title: A Phase II Study To Assess The Efficacy of Amifostine for Submandibular and Sublingual Salivary Sparing During Head and Neck Cancer Treatment With Intensity- Modulated Radiation Therapy (IMRT) for Parotid Salivary Sparing
Brief Title: Amifostine With IMRT for Submandibular and Sublingual Salivary Sparing During Head and Neck Cancer Treatment
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Study terminated by Principal Investigator; no patients completed study.
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: MedImmune LLC (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2006-0234
Record Dates: First submitted 2006-12-07; First posted 2006-12-08 (Estimated); Results first posted 2010-01-18 (Estimated); Last update posted 2012-08-07 (Estimated); Status verified 2012-07

CONDITIONS: Head and Neck Cancer
Keywords: Head and Neck Cancer; HNSCC; Submandibular and Sublingual Salivary Sparing; Amifostine; Ethyol; Radiation Therapy
MeSH Terms: conditions — Head and Neck Neoplasms; Squamous Cell Carcinoma of Head and Neck | interventions — Amifostine; Radiotherapy, Intensity-Modulated

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- IMRT + Amifostine (Experimental): Intensity-Modulated Radiation Therapy (IMRT) 2.0 to 2.2 Gy delivered in 30 fractions + Amifostine 500 mg, 2 divided doses subcutaneously 30-60 minutes prior to IMRT.
  Interventions: Drug: Amifostine; Procedure: Intensity- Modulated Radiation Therapy

INTERVENTIONS:
Drug: Amifostine — 500 mg in two divided doses subcutaneously given 30-60 minutes prior to IMRT.
  Other Names: Ethyol
Procedure: Intensity- Modulated Radiation Therapy — 2.0 to 2.2 Gy delivered in 30 fractions
  Other Names: IMRT

SUMMARY:
Primary Objective:

To determine if amifostine in combination with IMRT can mitigate the decrease in production of saliva by the submandibular and sublingual salivary glands in patients with HNSCC.

Secondary Objectives:

1. To establish a parotid gland dose volume histogram (DVH) versus measured flow relationship in this patient population:

   * When the mean dose is < 24-26 Gy (shift recovery time to left)
   * When the mean dose is > 24-26 Gy (DVH shift)
2. To observe mucositis in the following lower dose RT areas:

   * Upper lip
   * Lower lip
   * Right cheek
   * Left cheek
   * Right ventral and lateral tongue
   * Left ventral and lateral tongue
   * Floor of the mouth
   * Soft palate
   * Hard palate.
3. To observe the incidence and patterns of occipital scalp epilation;
4. To observe the incidence of dysphagia using the List Performance Status Scale (LPSS); and
5. To further evaluate the safety profile of amifostine in this patient population.

DETAILED DESCRIPTION:
Amifostine is designed to protect the cells in normal tissues against the toxicities of chemotherapy and radiation therapy.

Before you can start treatment on this study, you will have "screening tests." These tests will help the doctor decide if you are eligible to take part in this study.

Blood (about 2 tablespoons) will be drawn for routine blood tests. Your complete medical history will be recorded. You will have a physical exam, including measurement of your vital signs (blood pressure, heart rate, temperature, and breathing rate), weight, and height. You will have a dental exam. You will complete a questionnaire that asks questions about dry mouth. In addition, you will be asked questions about your diet and eating habits. This should take no longer than 10 minutes. Also, saliva will be collected by a simple, in-office oral test that measures saliva flow rate over a 5 minute period. Women who are able to have children must have a negative blood (about 1-2 teaspoons) pregnancy test.

If you are found to be eligible to take part in this study, you will receive IMRT Monday -Friday over a 6-7 week period. In addition, 2-3 hours before IMRT, you will also take pre-medications by mouth to prevent potential nausea and skin reactions (anti-nausea & antihistamine), including drinking water.You will receive daily IMRT therapy, excluding weekends and holidays. The radiation dose is designed to conform to the 3-dimensional shape of the tumor by controlling the intensity of the radiation beam to focus a higher radiation dose on the tumor (and not the surrounding normal tissue). Thirty (30) to 60 minutes before every IMRT treatment, you will receive study drug in two injections beneath the skin. IMRT will take about 30 minutes to complete.

Every day that you are receiving IMRT (Monday-Friday), you will be asked about any drugs you are taking and any side effects you are experiencing. Your vital signs will be recorded.

Every week (Weeks 2-7), you will have a complete oral and physical exam. You will complete the questionnaire that asks questions about dry mouth. You will be asked questions about your ability to perform daily activities (performance status evaluation). Your weight will also be measured. You will be asked to complete the symptom survey (the M.D. Anderson Symptom Inventory) that will ask you to rate your symptoms and how much the symptoms interfere in your daily activities.

On the last day you receive IMRT or amifostine (whichever is last), you will have a complete oral exam and you will complete the questionnaire about dry mouth.

Six (6) weeks after the end of therapy, you will have an end-of-therapy visit. At this visit, you will have a complete physical and oral exam with a saliva collection. You will complete the questionnaire about dry mouth. Your weight will be measured, and you will have a performance status evaluation. Blood (about (2) tablespoons) will be drawn for routine blood tests. You will be asked about any drugs you are taking and any side effects you are experiencing. In addition, you will be asked questions about your diet and eating habits.

You will be asked to complete the symptom survey (the M.D. Anderson Symptom Inventory) that will ask you to rate your symptoms and how much the symptoms interfere in your daily activities every week for 2 months after the end of radiation therapy. After this point, you will be asked to complete the symptom survey every month for 1 year.

You will have follow-up visits 4, 7, 10, and 12 months after the end of therapy. At these visits, you will have a complete oral exam and saliva collection. You will complete the dry mouth questionnaire. Your weight will be measured, and you will have a performance status evaluation and you will be asked questions about your diet and eating habits.

THIS IS AN INVESTIGATIONAL STUDY. Amifostine is FDA approved and commercially available. Amifostine is FDA approved to be given through a needle in your vein but not FDA approved to be given through a needle under the skin.

Up to 20 patients will take part in this study. All patients will be enrolled at M. D. Anderson.

ELIGIBILITY:
Inclusion Criteria:

1. Adult men and women of at least 18 years of age at the time of patient entry;
2. Women of reproductive potential (defined as being <1 year post-menopausal) must have a negative serum pregnancy test within 7 days of study entry;
3. Men and women of reproductive potential must agree to practice an effective method of avoiding pregnancy (including oral or implanted contraceptives, intrauterine device (IUD), female condom, diaphragm with spermicide, cervical cap, use of a condom by the sexual partner or sterile sexual partner) beginning at the time the informed consent is signed, and must agree to continue using such precautions while receiving IMRT through 6 weeks after the last dose of amifostine or RT, whichever is the last therapy discontinued;
4. Patients undergoing definitive or post-operative IMRT as follows:
5. Definitive Patients: Histology confirmed unknown primary T0N1-2bM0 or oropharynx Stage I, II, III, IV (TX, T1-T2, favorable T3 (exophytic) N0-N2b, M0), small volume primary and nodal, not requiring chemotherapy during RT (i.e., induction chemo is acceptable as well as concurrent biological therapy e.g., Cetuximab), squamous cell carcinoma (AJCC Staging of HNSCC). Lymph nodes bilaterally of the neck are at risk for metastatic disease and require irradiation per clinical judgment.
6. Post-operative Patients: Histology confirmed oral cavity, oropharynx, larynx and hypopharynx squamous cell carcinoma (AJCC Staging of HNSCC): *Stage III and IV squamous cell carcinoma treated with surgery as the primary modality requiring post-operative RT, but not receiving concurrent chemotherapy. *Indications for post-operative RT include: unfavorable T3 and T4 primaries, compromised margins, nodal metastases, extracapsular nodal extension, perineural invasion and lymphovascular invasion.
7. Zubrod performance status of 0 or 1
8. Adequate nutritional status as determined by the treating physician in conjunction with consultation with clinical nutritionists, as indicated.
9. Hemoglobin must be greater than or equal to 10 g/dL.
10. At least one parotid should keep a mean RT dose of < 24-26 Gy. If this cannot be achieved on one side, then the contralateral parotid dosing goal is to keep the mean dose as low as possible, typically <15 Gy.
11. It is anticipated that at least one submandibular gland will receive a mean dose >24-26 Gy.
12. Written informed consent and HIPAA authorization obtained from the patient prior to receipt of any study medication or beginning study procedures.

Exclusion Criteria:

1. Evidence of significant wound infection, fistula, or major wound dehiscence at time of patient entry.
2. Carcinomas of the paranasal sinuses, nasopharynx, or N3 at time of patient entry.
3. Presence of prior malignancies <5 years other than non-melanoma skin cancer or cervical, breast or bladder cancer in situ.
4. T3N0 glottic cancer at time of patient entry.
5. Prior chemotherapy for other cancer within less than or equal to 3 years prior to patient entry.
6. Planned concurrent or adjuvant chemotherapy.
7. Less than gross total resection for patients on post-operative RT.
8. Prior head neck irradiation except for localized non-melanomatous cutaneous carcinomas.
9. Salivary gland disease, e.g. Sjogren's disease at time of patient entry.
10. Pregnant or nursing at the time of patient entry or positive serum pregnancy test within 7 days of study entry.
11. Use of pilocarpine or cevimeline during participation in the study.
12. General medical or psychological conditions that might preclude the patient from completion of the study or from understanding and signing the informed consent.
13. Evidence of distant metastases.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2006-12; Primary Completion 2009-01 (Actual); Study Completion 2009-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mark Chambers, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- U.T. M.D. Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: Related Info — http://www.mdanderson.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment Period: 06/12/07 through 01/14/08. All participants recruited at UT MD Anderson Cancer Center.
Pre-assignment Details: Study terminated due to slow accrual and change in sponsor. Three patients registered, two removed prior to study beginning as not eligible.
Period: Overall Study
Arm/Group | IMRT + Amifostine
Started | 1
Completed | 0
Not Completed | 1
Not completed — Physician Decision | 1

BASELINE CHARACTERISTICS:
Arm/Group | IMRT + Amifostine
Number analyzed (Participants) | 1
Age Continuous [Median (Full Range); unit: years] | 48 [48 to 48]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 1
Region of Enrollment [Number; unit: participants]
  United States | 1

OUTCOME MEASURES:

1. Primary Outcome: 12-month Clinically Relevant Salivary Flow (CRSF)
Description: Primary endpoint is bilateral, 12-month Clinically Relevant Salivary Flow (CRSF) by the submandibular and sublingual salivary glands, collectively. Saliva production will be quantified using selective quantitative submandibular sialometry (total collection time of 5 minutes). A CRSF is equivalent to production of 0.05 mL of saliva post-radiation in a 5-minute collection period.
Time Frame: 12 months
Population: No analysis performed; study terminated early due to change in sponsor.
Arm/Group | IMRT + Amifostine
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: 1 year, 8 months
Description: No analysis done study terminated early. No patients completed study.
Arm/Group | IMRT + Amifostine
Serious Adverse Events (participants affected / at risk) | 0/0
Other Adverse Events (participants affected / at risk) | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No